CLINICAL TRIAL: NCT02621710
Title: Goal Achievement and Patient Satisfaction in Benign Hysterectomy
Status: Completed | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Graham Chapman, Resident, University Hospitals Cleveland Medical Center
Other Study IDs: 053161
Record Dates: First submitted 2015-11-28; First posted 2015-12-03 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Hysterectomy; Goal Achievement; Patient Satisfaction; Minimally Invasive Surgery
MeSH Terms: conditions — Patient Satisfaction | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Minimally invasive hysterectomy: Patients undergoing scheduled minimally invasive hysterectomy (vaginal, laparoscopic, robotic) for benign condition
  Interventions: Other: Questionnaire 3 months post-operatively
- Abdominal hysterectomy: Patients undergoing scheduled abdominal hysterectomy for benign condition
  Interventions: Other: Questionnaire 3 months post-operatively

INTERVENTIONS:
Other: Questionnaire 3 months post-operatively

SUMMARY:
This study evaluates patient goal achievement and satisfaction in benign hysterectomy. Patient's will state their goals prior to undergoing benign hysterectomy, and will receive a follow-up questionnaire 3 months post-operatively evaluating their perception of goal achievement and overall satisfaction. Goal achievement and satisfaction will be evaluated for association with surgical indication, surgical approach (minimally invasive vs abdominal surgery), and demographic information.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing hysterectomy for benign indication
* Age 18 or greater
* English speaking
* Access to communication via telephone

Exclusion Criteria:

* Patient undergoing hysterectomy for malignant or pre-malignant condition
* Non-english speaking patient
* Patient without telephone access
* Patient undergoing emergent or unplanned hysterectomy
* Vulnerable populations

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing benign hysterectomy for benign indications in a scheduled manner
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2015-12; Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Goal achievement score of 4 or 5 | 3 months post-operatively
  Patients will state their goals prior to surgery, then at the three months post-operatively will rank if their goals were met on a 1-5 likert scale (1=strongly disagree, 2=disagree, 3=neutral, 4=agree, 5=strongly agree). Goals are considered achieved with a likert score of 4 or 5.

SECONDARY OUTCOMES:
Percent of patient satisfaction | 3 months post-operatively
  At three months post-operatively, patients will state how satisfied they are with their hysterectomy experience, from 0 to 100%.

CONTACTS AND LOCATIONS:
Overall Officials: Sangeeta Mahajan, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals, Cleveland, Ohio, United States

REFERENCES:
- [Background] Pilzek AL, Raker CA, Sung VW. Are patients' personal goals achieved after pelvic reconstructive surgery? Int Urogynecol J. 2014 Mar;25(3):347-50. doi: 10.1007/s00192-013-2222-8. Epub 2013 Sep 18. PMID 24045936
- [Background] Mamik MM, Rogers RG, Qualls CR, Komesu YM. Goal attainment after treatment in patients with symptomatic pelvic organ prolapse. Am J Obstet Gynecol. 2013 Nov;209(5):488.e1-5. doi: 10.1016/j.ajog.2013.06.011. Epub 2013 Jun 13. PMID 23770473
- [Background] Hullfish KL, Bovbjerg VE, Gibson J, Steers WD. Patient-centered goals for pelvic floor dysfunction surgery: what is success, and is it achieved? Am J Obstet Gynecol. 2002 Jul;187(1):88-92. doi: 10.1067/mob.2002.124838. PMID 12114893
- [Background] Elkadry EA, Kenton KS, FitzGerald MP, Shott S, Brubaker L. Patient-selected goals: a new perspective on surgical outcome. Am J Obstet Gynecol. 2003 Dec;189(6):1551-7; discussion 1557-8. doi: 10.1016/s0002-9378(03)00932-3. PMID 14710061
- [Background] Mahajan ST, Elkadry EA, Kenton KS, Shott S, Brubaker L. Patient-centered surgical outcomes: the impact of goal achievement and urge incontinence on patient satisfaction one year after surgery. Am J Obstet Gynecol. 2006 Mar;194(3):722-8. doi: 10.1016/j.ajog.2005.08.043. PMID 16522404
- [Background] Nieboer TE, Johnson N, Lethaby A, Tavender E, Curr E, Garry R, van Voorst S, Mol BW, Kluivers KB. Surgical approach to hysterectomy for benign gynaecological disease. Cochrane Database Syst Rev. 2009 Jul 8;(3):CD003677. doi: 10.1002/14651858.CD003677.pub4. PMID 19588344
- [Background] ACOG Committee Opinion No. 444: choosing the route of hysterectomy for benign disease. Obstet Gynecol. 2009 Nov;114(5):1156-1158. doi: 10.1097/AOG.0b013e3181c33c72. PMID 20168127
- [Background] Martino MA, Berger EA, McFetridge JT, Shubella J, Gosciniak G, Wejkszner T, Kainz GF, Patriarco J, Thomas MB, Boulay R. A comparison of quality outcome measures in patients having a hysterectomy for benign disease: robotic vs. non-robotic approaches. J Minim Invasive Gynecol. 2014 May-Jun;21(3):389-93. doi: 10.1016/j.jmig.2013.10.008. Epub 2013 Oct 26. PMID 24513969
- [Background] Warren L, Ladapo JA, Borah BJ, Gunnarsson CL. Open abdominal versus laparoscopic and vaginal hysterectomy: analysis of a large United States payer measuring quality and cost of care. J Minim Invasive Gynecol. 2009 Sep-Oct;16(5):581-8. doi: 10.1016/j.jmig.2009.06.018. PMID 19835801
- [Background] Wright KN, Jonsdottir GM, Jorgensen S, Shah N, Einarsson JI. Costs and outcomes of abdominal, vaginal, laparoscopic and robotic hysterectomies. JSLS. 2012 Oct-Dec;16(4):519-24. doi: 10.4293/108680812X13462882736736. PMID 23484557
- [Background] Pitter MC, Simmonds C, Seshadri-Kreaden U, Hubert HB. The impact of different surgical modalities for hysterectomy on satisfaction and patient reported outcomes. Interact J Med Res. 2014 Jul 17;3(3):e11. doi: 10.2196/ijmr.3160. PMID 25048103